CLINICAL TRIAL: NCT02040584
Title: A Multicentre, Randomised, Open-label, Controlled, 12-month Follow-up Study to Assess Impact on Renal Function of an Immunosuppression Regimen Based on Tacrolimus Minimisation in Association With Everolimus in de Novo Liver Transplant Recipients. The REDUCE Study.
Brief Title: A Multicentre, Randomised, Open-label, Controlled, 12-month Follow-up Study to Assess Impact on Renal Function of an Immunosuppression Regimen Based on Tacrolimus Minimisation in Association With Everolimus in de Novo Liver Transplant Recipients.
Acronym: REDUCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001HES01; 2013-001191-38 (EudraCT Number)
Record Dates: First submitted 2014-01-07; First posted 2014-01-20 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-03

CONDITIONS: Liver Transplant
Keywords: De Novo Liver Transplant, Tacrolimus Minimisation, Everolimus, Renal Function, Liver transplant, allograft rejection, xenograft rejection, host vs graft disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: A multicentre, randomized, open-label, controlled, exploratory clinical trial with 12-months (52 weeks) of follow-up".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimisation of TAC (Experimental): Treatment with rTAC+EVR+corticosteroids
  Interventions: Drug: Minimisation of TAC
- TAC + MMF + corticosteroids (Active Comparator): Treatment with TAC + MMF + corticosteroids
  Interventions: Drug: TAC + MMF + corticosteroids

INTERVENTIONS:
Drug: Minimisation of TAC — •EVR: Treatment started at a total daily dose of 2 mg within 24 hours after randomisation. The dose of EVR was adjusted upon reaching trough levels (C-0h) in whole blood of 3-8 ng/mL. The daily dose (in two administrations) of EVR may have been modified to maintain trough levels (C-0h) in whole blood of 3-8 ng/mL until Week 52 post-transplant. •TAC: Once confirmation was obtained, beginning in Week 5, that trough levels (C-0h) in whole blood of EVR were between 3-8 ng/mL, minimisation of TAC began, in order to reach trough levels (C-0h) of TAC in whole blood of ≤5 ng/mL no later than four weeks after randomisation (Week 8), which were levels that should have been maintained until Week 52 post-transplant. •MMF was withdrawn at the same time that EVR was introduced. •oral corticosteroids was administered in accordance with local clinical practice, although a therapeutic strategy free of corticosteroids was permitted
  Arms: Minimisation of TAC
Drug: TAC + MMF + corticosteroids — •Dose of TAC: Trough levels (C-0h) of TAC in whole blood should have been maintained between 6-10 ng/mL until Week 52 post-transplant. •Dose of MMF: Doses of 500-1000 mg/12 hrs was maintained until Week 52. •Corticosteroids: During the study, oral corticosteroids was administered in accordance with local clinical practice, although a therapeutic strategy free of corticosteroids was permitted (e.g. in patients with a history of HCV). It was recommended in any case that corticosteroids not be administered beyond Week 24 post-transplant except in cases of hepatopathy of autoimmune origin. At each centre all patients should have followed the same administration protocol for corticosteroids based on history of HCV.
  Arms: TAC + MMF + corticosteroids

SUMMARY:
Assuming greater efficacy in the prevention of acute rejection in the EVR arm with minimisation of TAC levels, the hypothesis of the present trial was that the introduction of EVR in combination with the minimisation of TAC (rTAC) may offer improved kidney function compared with standard therapy with TAC-MMF.

DETAILED DESCRIPTION:
A multicentre, randomized, open-label, controlled, exploratory clinical trial with 12-months (52 weeks) of follow-up.

ELIGIBILITY:
Screening Visit - Inclusion Criteria

1. Recipients age 18 or over receiving a first liver transplant from a cadaver donor.
2. Patients diagnosed with HCC must meet the Milan radiological criteria at the time of transplant (1 nodule ≤5 cm in diameter, or 2-3 nodules, all <3 cm in diameter) - at time of patient's inclusion on the waiting list.

   Anh: done.
3. Patients who have signed the informed consent to participate in the study.
4. Patients who by medical criteria are capable of complying with the study regimen.

Screening Visit - Exclusion Criteria

1. Recipients who have received multiple transplants of solid organs or pancreatic islet cells.
2. Patients who have previously received an organ or tissue transplant.
3. Patients with a combined liver-kidney transplant.
4. Recipients of lobes or segments of liver from a live donor.
5. A history of malignancy of any organ system in the previous 3 years according to local protocols (regardless of signs of local recurrence or metastasis), other than non-metastasising basal cell carcinoma or squamous cell carcinoma (epidermoid carcinoma) of the skin, or HCC.
6. Patients with known hypersensitivity to the drugs used in the study or others of their class, or to any of their excipients.
7. Recipients of ABO-incompatible transplants.
8. Patients who test positive for HIV.
9. Recipients of organs from donors who tested positive for the hepatitis B surface antigen or HIV seropositive.
10. Patients with any medical or surgical condition that in the opinion of the investigator may significantly alter the absorption, distribution, metabolism or excretion of the study medication.
11. Women of childbearing potential (i.e. women who are not postmenopausal with amenorrhoea of more than 1 year or surgically sterile) who are planning to become pregnant, are pregnant and/or breastfeeding, or who do not wish to use effective contraception, e.g. hormonal contraceptives (implantation, patches, oral) and double-barrier methods (any double combination of: IUD, male or female condoms with spermicidal gel, diaphragm, contraceptive sponge, cervical cap).
12. Patients who are taking part in another clinical trial.

Randomisation Visit - Inclusion Criteria

1. Functioning allograft at the time of randomisation. A functioning allograft is defined as:

   1. levels of AST, ALT and total bilirubin ≤ 4 times the upper limit of normal, and
   2. levels of alkaline phosphatase and GGT ≤ 5 times the upper limit of normal.
2. Glomerular filtrate ≥30 mL/min/1.73 m2 (calculated using the MDRD-4 equation).

Randomisation Visit - Exclusion Criteria

1. Patients with proteinuria ≥1.0 g/24 hrs confirmed in the urine sample (protein/creatinine ratio) that cannot be explained by immediate post-operative causes.
2. Patients with severe hypercholesterolaemia (≥350 mg/dL; ≥9 mmol/L) or severe hypertriglyceridaemia (≥750 mg/dL; ≥8.5 mmol/L).
3. Patients with a platelet count ≤50,000/mm3.
4. Patients with an absolute neutrophil count ≤1,000/mm3 or WBC count ≤2,000/mm3.
5. Patients who cannot take oral medication.
6. Patients with clinically significant systemic infection who require active use of intravenous antibiotics.
7. Patients who are in intensive care units and require vital support measures such as mechanical ventilation, dialysis, or vasoactive drugs.
8. Patients who have required renal replacement therapy in the 7 days prior to randomisation.
9. Patients who have had an episode of acute rejection and have required antibody therapy or who have had more than one episode of corticosteroid-sensitive acute rejection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2016-02-10 (Actual); Study Completion 2016-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- Spain (16):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barakaldo, Basque Country
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Santa Cruz de Tenerife
  - Novartis Investigative Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled were 217, patients in the safety population were 215, and patients in the ITT population were 211.
Pre-assignment Details: The intention-to-treat population (ITT) that was used for all efficacy analyses included all randomised patients who had received at least one dose of the study medication (safety population) and had at least one assessment subsequent to the randomisation visit for determining the primary efficacy endpoint.
Groups:
- Experimental Group: Minimisation of TAC: Treatment with rTAC+EVR+corticosteroids
- Control Group: Treatment with TAC + MMF + corticosteroids
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 105 | 106
Completed | 70 | 74
Not Completed | 35 | 32
Not completed — Adverse Event | 13 | 6
Not completed — Protocol Violation | 9 | 11
Not completed — Unsatisfactory therapeutic effect | 0 | 1
Not completed — Death | 6 | 3
Not completed — Transplant rejection/retransplant | 0 | 1
Not completed — Immunosuppressant/prohibited med use | 7 | 10

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomised patients who had received at least one dose of the study medication and had at least one assessment subsequent to the randomization visit for determining the primary efficacy endpoint. Patients were analysed according to the treatment to which they were assigned at randomisation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 105 | 106 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.43 (6.37) | 55.84 (7.45) | 57.13 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 91 | 90 | 181

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Participants Showing Clinical Benefit by Renal Function Stratification
Description: Clinical benefit is defined as: • an improvement in 1 or 2 ranges of the eGFR, according to MDRD-4 at Week 52 post-transplant in patients with values of 30-<45 or 45-<60 mL/min/1.73 m2 in Week 4. or • stabilisation of eGFR in patients with values ≥60 mL/min/1.73 m2 at Week 4 and maintained at Week 52 post-transplant.
Time Frame: week 4, week 52.
Population: ITT
Measure: Number; unit: Percentages of partcipants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 105 | 106
Percentages of partcipants
  > = 30 - 45 ml/min/1.73m^2 at Week 52 | 4.76 | 3.77
  > = 45 - <60 ml/min/1.73m^2 at Week 52 | 14.29 | 16.04
  > = 60 ml/min/1.73m^2 at Week 52 | 79.05 | 79.25
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Null hypothesis (H0): there were no differences in kidney function between the two groups, in contrast with the alternative hypothesis (H1), in which there were differences: HO: CBS = CBC versus H1: CBS ≠ CBC, where CBS and CBC were percentages of patients who showed clinical benefit at Week 52 for the study group and control group, respectively; Test type: Superiority or Other; p = 0.9423, Fisher Exact; Week 52

2. Secondary Outcome: Changes in Creatinine Clearance - Cockcroft-Gault Formula
Description: Kidney function was assessed over time by creatine clearance based on the Cockcroft-Gault formula.
  Estimated creatinine clearance (mL/min) = [(140 - age) x (weight) x (0.85 if female)] / (72 x serum creatinine).
  Units: age (years); weight (kg); serum creatinine (mg/dL). The values of the eGFR according to the creatinine clearance (Cockcroft-Gault formula) for the ITT population were ml/min/1.73 m^2.
Time Frame: Screening visit (transplant), weeks 1,4,12,24,36 and 52 post-transplant
Population: ITT
Measure: Mean (Standard Deviation); unit: ml/min/1.73m^2
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 105 | 106
ml/min/1.73m^2
  Screening | 104.67 (36.40) | 109.69 (48.47)
  Week 1 | 116.93 (44.82) | 118.09 (44.82)
  Week 4 | 80.19 (28.00) | 91.26 (37.60)
  Week 12 | 87.76 (26.51) | 90.14 (35.82)
  Week 24 | 89.57 (32.89) | 87.93 (35.92)
  Week 36 | 94.46 (30.26) | 90.91 (35.96)
  Week 52 | 92.21 (29.96) | 91.04 (37.26)

3. Secondary Outcome: Changes in eGFR Based on the MDRD-4 Formula
Description: Kidney function was assessed over time by changes in eGFR according to the MDRD-4 formula. The MDRD-4 formula (Levey et al., 2000) was used based on serum concentration of creatinine (conventional units): eGFR (mL/min/1.73 m2) = 186 x (serum creatinine)-1.154 x (age)-0.203 x (0.742 if female) x (1.210 if of African descent).
  Units: serum creatinine (mg/dL); age (years).
Time Frame: Screening visit (transplant), weeks 1,4,12,24,36 and 52 post-transplant
Population: ITT
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 105 | 106
ml/min/1.73m2
  Screening | 100.20 (38.74) | 99.42 (43.09)
  Week 1 | 112.86 (50.06) | 112.15 (48.16)
  Week 4 | 82.18 (28.47) | 88.39 (34.32)
  Week 12 | 85.99 (25.13) | 83.57 (28.19)
  Week 24 | 86.02 (31.97) | 82.00 (26.93)
  Week 36 | 87.68 (32.49) | 83.04 (25.56)
  Week 52 | 86.09 (27.87) | 83.23 (25.24)

4. Secondary Outcome: eGFR Values(MDRD-4 Formula) According to the MELD Score
Description: Model for End Stage Liver Disease (MELD) score: ≤14, 15-19, 20-24, 25-29, ≥30. The higher the number indicates the urgency for transplant.
Time Frame: Screening visit (transplant), weeks 1,4,12,24,36 and 52 post-transplant
Population: ITT population (patients with MDRD-4 values).
Measure: Median (Inter-Quartile Range); unit: ml/min/1.73m^2
Groups:
- <= 14: Experimental group (Minimisation of TAC: Treatment with rTAC+EVR+corticosteroids) with MELD score <= 14
- 15 to 19: Experimental group (Minimisation of TAC: Treatment with rTAC+EVR+corticosteroids) with MELD score 15-19
- 20 to 24: Experimental group (Minimisation of TAC: Treatment with rTAC+EVR+corticosteroids) with MELD score 20 to 24
- 25 to 29: Experimental group (Minimisation of TAC: Treatment with rTAC+EVR+corticosteroids) with MELD score 25 to 29
- > = 30: Experimental group (Minimisation of TAC: Treatment with rTAC+EVR+corticosteroids) with MELD score > = 30
- <= 14 Control Group: Control group (Treatment with TAC + MMF + corticosteroids) with MELD score <= 14
- 15 to 19 Control Group: Control group (Treatment with TAC + MMF + corticosteroids) with MELD score 15 to 19
- 20 to 24 Control Group: Control group (Treatment with TAC + MMF + corticosteroids) with MELD score 20 to 24
- 25 to 29 Control Group: Control group (Treatment with TAC + MMF + corticosteroids) with MELD score 25 to 29
- > = 30 Control Group: Control group (Treatment with TAC + MMF + corticosteroids) with MELD score > = 30
Arm/Group | <= 14 | 15 to 19 | 20 to 24 | 25 to 29 | > = 30 | <= 14 Control Group | 15 to 19 Control Group | 20 to 24 Control Group | 25 to 29 Control Group | > = 30 Control Group
Number analyzed (Participants) | 52 | 25 | 21 | 5 | 1 | 56 | 24 | 18 | 3 | 4
ml/min/1.73m^2
  Screening | 96.63 [76.31 to 119.50] | 90.29 [65.64 to 114.92] | 88.89 [70.03 to 114.67] | 104.45 [93.21 to 123.90] | 38.35 [38.35 to 38.35] | 102.27 [75.09 to 120.19] | 93.85 [73.93 to 123.19] | 91.45 [68.74 to 116.49] | 99.50 [19.76 to 137.89] | 53.73 [38.82 to 66.97]
  Week 1 | 114.00 [94.24 to 142.51] | 93.31 [76.61 to 127.75] | 83.45 [66.76 to 114.06] | 137.61 [124.30 to 148.67] | 82.04 [82.04 to 82.04] | 108.64 [83.22 to 138.55] | 92.98 [55.41 to 129.49] | 119.19 [100.53 to 147.60] | 156.41 [29.81 to 184.87] | 86.45 [57.98 to 117.96]
  Week 4 | 81.37 [63.46 to 92.20] | 85.19 [66.09 to 99.26] | 70.57 [51.90 to 99.02] | 75.94 [50.93 to 121.86] | 69.43 [69.43 to 69.43] | 89.44 [62.78 to 107.55] | 72.76 [51.64 to 113.93] | 89.67 [63.89 to 133.44] | 85.23 [42.83 to 109.13] | 78.57 [51.47 to 108.61]
  Week 12 | 85.81 [64.65 to 98.87] | 88.76 [65.92 to 118.20] | 83.91 [68.46 to 94.96] | 94.82 [50.94 to 106.28] | 56.67 [56.67 to 56.67] | 83.63 [69.33 to 101.35] | 67.00 [48.31 to 99.84] | 87.22 [67.63 to 107.01] | 65.01 [43.15 to 96.53] | 81.92 [58.33 to 87.43]
  Week 24 | 80.76 [64.37 to 107.89] | 81.41 [57.22 to 104.86] | 78.88 [62.22 to 94.68] | 84.86 [68.54 to 101.19] | 60.37 [60.37 to 60.37] | 80.01 [66.16 to 97.47] | 70.27 [55.26 to 93.99] | 82.64 [65.25 to 113.80] | 88.34 [30.17 to 104.72] | 62.74 [47.46 to 75.65]
  Week 36 | 81.96 [64.82 to 111.44] | 92.44 [68.05 to 113.18] | 75.62 [61.64 to 100.46] | 83.09 [55.72 to 110.46] | 58.07 [58.07 to 58.07] | 86.72 [72.09 to 97.40] | 67.90 [54.34 to 90.95] | 86.17 [68.59 to 107.21] | 68.32 [57.01 to 79.63] | 65.58 [45.11 to 73.55]
  Week 52 | 86.14 [66.70 to 101.59] | 88.94 [65.24 to 114.50] | 71.60 [62.48 to 89.66] | 83.94 [60.69 to 107.20] | 53.93 [53.93 to 53.93] | 80.92 [68.98 to 104.03] | 70.32 [54.12 to 82.38] | 90.66 [74.52 to 113.18] | 74.82 [69.00 to 80.63] | 63.26 [45.52 to 79.77]

5. Secondary Outcome: Urine Protein/Creatinine Ratio
Description: The urine protein/creatinine ratio was assessed throughout follow-up in both treatment groups.
Time Frame: Screening visit, week 1,4,18,24, and 52
Population: ITT
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 105 | 106
mg/g
  Screening | 199.89 (582.03) | 131.56 (178.95)
  Week 1 | 252.48 (308.22) | 349.46 (396.44)
  Week 4 | 134.77 (175.05) | 141.71 (187.11)
  Week 18 | 204.26 (688.05) | 105.02 (79.61)
  Week 24 | 200.17 (466.55) | 120.52 (108.04)
  Week 52 | 219.41 (406.52) | 143.05 (220.72)

6. Secondary Outcome: Percentage of Participants With Incidence of Proteinuria
Description: The incidence of proteinuria (≥0.5-0.9 g/day, ≥1.0-2.9 g/day and ≥3.0 g/day) was assessed throughout follow-up in both treatment groups. Proteinuria was defined as protein/creatinine ratio ≥ 0.5.
Time Frame: Screening visit, week 1,4,18,24, and 52
Population: ITT
Measure: Number; unit: Percentages of participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 105 | 106
Percentages of participants
  ≥ 0.5-1.0 g/day at screening | 0.00 | 3.77
  ≥ 1.0-3.0 g/day at screening | 2.00 | 1.89
  ≥ 3.0 g/day at screening | 2.00 | 0.00
  ≥ 0.5-1.0 g/day at Week 1 | 3.23 | 18.31
  ≥ 1.0-3.0 g/day at Week 1 | 6.45 | 5.63
  ≥ 3.0 g/day at Week 1 | 0.00 | 0.00
  ≥ 0.5-1.0 g/day at Week 4 | 5.21 | 1.05
  ≥ 1.0-3.0 g/day at Week 4 | 0.00 | 1.05
  ≥ 3.0 g/day at Week 4 | 0.00 | 0.00
  ≥ 0.5-1.0 g/day at Week 18 | 0.00 | 0.00
  ≥ 1.0-3.0 g/day at Week 18 | 1.39 | 0.00
  ≥ 3.0 g/day at Week 18 | 1.39 | 0.00
  ≥ 0.5-1.0 g/day at Week 24 | 7.58 | 1.52
  ≥ 1.0-3.0 g/day at Week 24 | 0.00 | 0.00
  ≥ 3.0 g/day at Week 24 | 1.52 | 0.00
  ≥ 0.5-1.0 g/day at Week 52 | 6.67 | 1.89
  ≥ 1.0-3.0 g/day at Week 52 | 3.33 | 1.89
  ≥ 3.0 g/day at Week 52 | 0.00 | 0.00

7. Secondary Outcome: Percentage of Participants With Acute Rejection, BPAR, and Treated BPAR
Description: Liver biopsy had to be performed in all cases where acute rejection was suspected. Results of the biopsy were interpreted by the local pathologist (who did not known the treatment given to the patient) according to the Banff classification (1997).
  Biopsy-proven acute rejection (BPAR) defined as clinical suspicion of acute rejection confirmed in biopsy.
  Treated BPAR was deemed to be an episode of acute rejection in which the interpretation of the local pathologist showed that it reached any grade of acute rejection under the Banff classification, and for which anti-rejection therapy was administered.
  Loss of the liver allograft was deemed to have occurred the day that the patient was again included on the waiting list for liver transplant, the day he or she received another allograft or upon the death of the patient.
  All suspected hepatic allograft rejections were considered acute rejection
Time Frame: Throughout the study period, approximately 2 years and 2 months
Population: ITT
Measure: Number; unit: Percentages of participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 105 | 106
Percentages of participants
  Patients with suspected acute rejection | 17.14 | 15.09
  Patients with BPAR | 5.71 | 3.77
  Patients with treated BPAR | 4.76 | 1.89

8. Secondary Outcome: Time to Rejection
Description: Time to acute rejection was calculated from the date of transplantation. Acute rejection date was taken from biopsy date, as the date of rejection was not collected.
  Time to treated BPAR was calculated from the date of transplantation.
Time Frame: Throughout study period, approximately 2 years and 2 months
Population: ITT
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 105 | 106
months
  Time to acute rejection | 3.74 (3.15) | 2.91 (2.89)
  Time to treated BPAR | 2.65 (1.50) | 3.85 (5.25)

9. Secondary Outcome: Severity of Rejection
Description: Severity of acute rejection and treated BPAR was graded according to Banff criteria.
  Grade of acute rejection according to Banff criteria: mild, moderate, severe.
Time Frame: Throughout study period, approximately 2 years and 2 months
Population: ITT
Measure: Number; unit: Percentages of participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 105 | 106
Percentages of participants
  Severity of acute rejection: Mild (Grade I) | 13.64 (3.15) | 11.11 (2.89)
  Severity of acute rejection: Moderate(Grade II) | 13.64 (1.50) | 5.56 (5.25)
  Severity of acute rejection: Severe(Grade III) | 0.00 | 5.56
  Severity of treated BPAR: Mild (Grade I) | 33.33 | 0.00
  Severity of treated BPAR: Moderate(Grade II) | 50.00 | 50.00
  Severity of treated BPAR: Severe(Grade III) | 0.00 | 50.00

10. Secondary Outcome: Percentages of Participants With HCV-positive and HCV Genotype
Description: The viral load of HCV-RNA and HCV genotype was assessed in HCV-positive patients.
  The term "genotype" was used to describe strains of HCV that vary but were related to the virus. Worldwide, there were 11 primary groups of HCV genotypes designated by the numbers from 1-11, with the most common in our setting being subtypes 1a, 1b, 2 and 3, which were identified in the local laboratory according to their usual testing methods.
Time Frame: approximately 2 years and 2 months
Population: ITT
Measure: Number; unit: Percentages of participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 105 | 106
Percentages of participants
  Hepatitis C virus (HVC) positive: number analyzed (Participants) | 35 | 39
  Hepatitis C virus (HVC) positive | 33.33 | 36.79
  HCV genotype 01: number analyzed (Participants) | 28 | 30
  HCV genotype 01 | 80.00 | 76.92
  HCV genotype 02: number analyzed (Participants) | 0 | 0
  HCV genotype 03: number analyzed (Participants) | 6 | 4
  HCV genotype 03 | 17.14 | 10.26
  HCV genotype 04: number analyzed (Participants) | 1 | 1
  HCV genotype 04 | 2.86 | 2.56
  HCV genotype 05: number analyzed (Participants) | 0 | 0
  HCV genotype 06: number analyzed (Participants) | 0 | 0
  HCV genotype 07: number analyzed (Participants) | 0 | 0
  non-responders: number analyzed (Participants) | 0 | 4
  non-responders |  | 10.26

11. Secondary Outcome: Concentration of p-P70S6K
Description: the biomarker of personal response to everolimus, monitoring of the activity of the target, kinase P70 S6, in its phosphorylated form at Thr389.
  EVR=everolimus Cmin=minimum concentration
Time Frame: weeks 6,8,12,18,24,36,52 at 0 (Cmin), and 1 (C1h) hrs post-dose.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Experimental Group
Number analyzed (Participants) | 74
ng/ml
  Cmin EVR week 6 | 3.8 (1.7)
  C1h EVR week 6 | 6.8 (6.3)
  Cmin EVR week 8 | 4.7 (1.6)
  C1h EVR week 8 | 9.5 (4.9)
  Cmin EVR week 12 | 4.4 (1.8)
  C1h EVR week 12 | 16 (9.5)
  Cmin EVR week 18 | 6.8 (2.7)
  C1h EVR week 18 | 14.6 (6.7)
  Cmin EVR week 24 | 5.3 (2.13)
  C1h EVR week 24 | 18 (7.2)
  Cmin EVR week 36 | 5.1 (1.35)
  C1h EVR week 36 | 12.7 (4.2)
  Cmin EVR week 52 | 5.35 (0.97)
  C1h EVR week 52 | 16.1 (7.6)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 2 years and 2 month.
Description: AE and SAE analyses were done on the safety population (N=215). The safety population included all randomised patients who had received at least one dose of the study medication. Patients were analysed according to the treatment received. All safety analyses were based on the safety population.
Arm/Group | Experimental Group | Control Group
Serious Adverse Events (participants affected / at risk) | 55/106 | 48/109
Other Adverse Events (participants affected / at risk) | 97/106 | 105/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group (N=106) | Control Group (N=109)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 1
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 6 | 3
Strangulated hernia (General disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 4 | 3
Bile duct stone (Hepatobiliary disorders) | 2 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Budd-Chiari syndrome (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 2 | 1
Cholestasis (Hepatobiliary disorders) | 2 | 3
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 | 1
Hepatic artery stenosis (Hepatobiliary disorders) | 1 | 0
Hepatic artery thrombosis (Hepatobiliary disorders) | 2 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic ischaemia (Hepatobiliary disorders) | 0 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Liver transplant rejection (Immune system disorders) | 2 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 0
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Fungaemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 6 | 4
Herpes virus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Herpes zoster disseminated (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 2 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pseudomonas bronchitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 5 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 2 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 1
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 | 2
Complications of transplanted liver (Injury, poisoning and procedural complications) | 3 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Liver graft loss (Injury, poisoning and procedural complications) | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 4 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 | 0
Biopsy liver (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Endoscopic retrograde cholangiopancreatography (Investigations) | 4 | 2
Laboratory test (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of thorax (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Device ineffective (Product Issues) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 2 | 3
Renal impairment (Renal and urinary disorders) | 1 | 1
Renal tubular disorder (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Testicular cyst (Reproductive system and breast disorders) | 1 | 0
Testicular disorder (Reproductive system and breast disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Bile duct stent removal (Surgical and medical procedures) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 2
Arterial stenosis (Vascular disorders) | 0 | 1
Arterial thrombosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 1
Steal syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group (N=106) | Control Group (N=109)
Anaemia (Blood and lymphatic system disorders) | 30 | 36
Leukocytosis (Blood and lymphatic system disorders) | 6 | 7
Leukopenia (Blood and lymphatic system disorders) | 14 | 10
Neutropenia (Blood and lymphatic system disorders) | 4 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 24 | 22
Abdominal pain (Gastrointestinal disorders) | 8 | 11
Abdominal pain upper (Gastrointestinal disorders) | 6 | 3
Ascites (Gastrointestinal disorders) | 24 | 17
Constipation (Gastrointestinal disorders) | 13 | 7
Diarrhoea (Gastrointestinal disorders) | 20 | 29
Ileus paralytic (Gastrointestinal disorders) | 2 | 8
Vomiting (Gastrointestinal disorders) | 7 | 14
Asthenia (General disorders) | 11 | 16
Oedema (General disorders) | 8 | 5
Oedema peripheral (General disorders) | 39 | 27
Pyrexia (General disorders) | 15 | 17
Cholestasis (Hepatobiliary disorders) | 22 | 19
Jaundice (Hepatobiliary disorders) | 2 | 6
Hepatitis C (Infections and infestations) | 6 | 4
Urinary tract infection (Infections and infestations) | 6 | 8
Transaminases increased (Investigations) | 9 | 6
Cell death (Metabolism and nutrition disorders) | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 4 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 13
Dyslipidaemia (Metabolism and nutrition disorders) | 11 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 16 | 17
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 13
Headache (Nervous system disorders) | 11 | 12
Tremor (Nervous system disorders) | 13 | 19
Anxiety (Psychiatric disorders) | 7 | 3
Insomnia (Psychiatric disorders) | 17 | 10
Acute kidney injury (Renal and urinary disorders) | 5 | 6
Proteinuria (Renal and urinary disorders) | 11 | 2
Renal failure (Renal and urinary disorders) | 12 | 16
Renal impairment (Renal and urinary disorders) | 9 | 16
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 8
Hypertension (Vascular disorders) | 24 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.